CLINICAL TRIAL: NCT00862173
Title: Gene-expression Profile as Predictor of Central Nervous System Metastasis Development in Non-small Cell Lung Cancer: a Prospective Study
Brief Title: Gene-expression Profiles in CNS-metastatic Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, DR. MYRNA CANDELARIA, Gene expression Profiles in CNS metastasic Non small Cell Lung Cancer, National Institute of Cancerología
Other Study IDs: 008/025/OMI
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Brain Disease; Metastasis; Lung Cancer
Keywords: Gene-expression profile; Central nervous system metastasis; Non-small-cell lung cancer
MeSH Terms: conditions — Brain Diseases; Neoplasm Metastasis; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — NSCLC Biopsy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with NSCLC with CNS Metastasis: Patients who developed CNS metastasis of NSCLC during the treatment.
- Patients with NSCLC without CNS Metastasis: Patients with NSCLC that does not develop CNS metastasis during the treatment.

SUMMARY:
Non small-cell lung cancer (NSCLC) accounts 85% of all lung cancer.The development of brain metastasis diminished life expectancy to less than one year with a median survival of less than three months. In NSCLC cancer, approximately 50% of patients with locally advanced disease develop brain metastasis at some time during the natural of disease. The central nervous system constitutes the first site of recurrence in 15 to 40% of these patients. Microarrays evaluate the diagnosis, treatment and prognosis of lung cancer.There are no studies that specifically evaluate the relationship between a genetic profile of NSCLC and metastasis to the CNS, with the purpose of distinguishing a subgroup of patients that will benefit of prophylactic treatment.What is the association between a genetic profile on NSCLC and the development of CNS metastasis.Obtaining a genetic profile from the primary NSCLC tumor cells, by using microarrays, we can predict the development of CNS metastasis arise a subgroup of patients that could benefit from prophylactic cranial radiation with which their quality of life and prognosis most probably will increase.Objective:Determine the association between a genetic profile from the primary tumor cells and the development of central nervous system metastasis in patients with non small-cell lung cancer.A genetic profile from the primary tumor cells are associated with the development of central nervous system metastasis in patients with NSCLC. A clinical, prospective, analytic, open, non randomized, prognostic and observational cohort with 66 patients with NSCLC who authorize a biopsy study from February, 2008 to December, 2012, INMEGEN institute will be in charge of performing the microarrays and the computer analysis in order to obtain the different genetic profiles that will be differentially expressed related with CNS metastasis risk profiles. Patients will be followed-up by means of the external consult of lung neoplasms. The statistical analysis will be performed using tests like Student's t or Mann-Whitney's U test. A multivariate analysis of logistic regression will be performed. Global survival time will be analyzed using Kaplan-Meier's technique and the comparison between groups will be performed with log-rank test. The adjustment for potential confusors will be performed using multivariate regression analysis. For result representation, we will use tables and graphs and pertinent measures will be taken to disclose the study.

DETAILED DESCRIPTION:
Brain metastases occur in 30-50% of lung adenocarcinoma (LAC) patients and confer a worse prognosis and quality of life. A better selection of in-risk patients through a more accurate biomarker could improve the benefit of prophylactic therapies. The aim of this prospective study was to determine a gene-expression profile of primary tumor associated with brain metastasis (BM) and to evaluate the overall survival (OS) in patients with advanced LAC.

Introduction.Lung cancer is the first cause of cancer death in the world. Eighty five percent of patients are diagnosed yearly with non-small cell lung cancer (NSCLC). Despite efforts, innovations, and progress in diagnosis and treatment of these patients, overall survival (OS) at 5 years of diagnosis is only 15%. The central nervous system (CNS) is a devastating and frequent site of metastasis development in NSCLC. The reported incidence of CNS metastasis in patients with NSCLC is 54% with an OS of <1 year after diagnosis. Age, clinical stage, gender, and initial treatment period are some of the reported with CNS metastasis development-related factors in patients with NSCLC. We recently described that high carcino-embryonic antigen (CEA) serum levels (>40 ng/dL) at diagnosis and adenocarcinoma histological type are independently associated with higher risk if brain metastasis development. However, due to their lack of specificity of all this reported factors, we are required to detect biomarkers to predict brain metastasis in patients with NSCLC with the objective to prevent their development.Metastasis process is complex it involves well-defined molecular-printed steps, as invasion, vascular intravasation, implantation and growing at the new specific organ. Higher motility, capacity for extracellular matrix degradation, immune system evasion, and adhesion at the new specific organ are some of the tumoral cell characteristics required to metastasize. In particular, molecular events for brain metastasis development from primary NSCLC even if no at al described, are currently well understood. Gene-expression microarray allow analyzing the expression changes of thousands of genes simultaneously, distinguishing the altered expression of neoplastic cell genes from normal tissue. Identification of biological patterns, pharmacological molecular targets, and biomarkers for prognosis and evaluation for therapeutic response, and even a more specific neoplasia classification are some of the results of gene-expression microarray studies in hematological, breast and NSCLC cancer. Determination of tobacco-smoke transcriptional changes in oncogenes and antioncogenes had been determined by the use microarray data. A gene-expression profile of 20 genes differentiates health lung tissue and lung cancer with higher specificity than histopathologic evaluation. Furthermore, gene-expression microarray studies had been developed for predicting survival and recurrence in early NSCLC stages for identification of patients who could have benefit of adjuvant therapy, with promising result.The objective of this study was to identify a gene-expression profile from primary lung adenocarcinoma related with brain metastasis, and to evaluate in a prospective manner their prognostic significance on survival in patients with advanced disease.Experimental Design These study used clinical, longitudinal, prospective, observational, and analytical cohort s with the selection of a nonprobabalistic-type sample.In a prospective manner, from January 2009 to June 2011, patients admitted to our Institute confirmed histologically confirmed stage IIIb and IV of LAC were eligible for study inclusion. Analyzed clinical variables comprised smoking history, gender, age, general condition and brain metastasis development. Primary tumor core-biopsy was performed prior to any treatment and snap-frozen. A single pathologist evaluated all tumors. Standard platinum-based chemotherapy was employed for all patients. All patients were submitted to Magnetic resonance imaging (RM) to evidence the presence or absence of brain metastasis (BM). During follow-up, we carried out Computed tomography (CT) of the brain stem for this purpose. Preliminary statistical analysis was performed utilizing the Student t, the Mann-Whitney U, the χ2, or the Fisher exact test. Once the study ends, we will conduct logistic-regression multivariate analysis. Global survival time will be analyzed with the Kaplan-Meier technique, and comparisons among groups will be performed with the log-rank test. High Risk characteristics as gender, histology, and age related with greater frequency of development of metastasis to CNS were analyzed.The study was carried out according to the principles of ClinicalTrials and accepted by the INCan Bioethical and Scientific Committees (reference numbers INCAN/CC/067/08). A collaboration agreement was signed with the INMEGEN and was approved within the Health Research Sectorial Fund (FSIS) CONACyT-México (SALUD-2009-01-115552).

Selection for obtaining tumor biopsies depended on the characteristics of the patient and of the tumor. The biopsy could be taken by means of CT guided tru-cut needle, open thoracoscopy, or bronchoscopy with optic fiber. Each tumor sample was divided into two; one sample was analyzed by the INCan Pathology Service (by a sole observer blinded to the clinical variables) for their histological clinical diagnosis and quantification of neoplastic cellularity, and the remaining half was immediately stored at -80°C until processing for RNA extraction.RNA Extraction:RNA was extracted from frozen tumor biopsies, weighted and cryofractured in liquid nitrogen. Extraction and purification of total RNA from tissue (up to 5 mg tissue) procedure was done using RNeasy Micro Kit (QIAGEN, Germany) (cat. 217084). RNA was analyzed using the Agilent 6000 Chip (Agilent Technologies, Santa Clara, C.A.). RNA quality consisted on the obtention of RNA Integrity Number (RIN) > 8. RNA samples were chosen for microarray analysis when quality and concentration were obtained for this purpose. Microarray Expression:We are using an Affymetrix platform, which consists of an in situ synthesized oligonucleotide microarray. The GeneChip® that we are employing is the Human Gene 1.0 ST Array, which allows analyzing the expression of 28,869 different genes (each transcript is represented by 26 disperse probes along its entire length, present in the human genome, which covers 99% of the sequences present in the RefSeq data bank of the GenBank. The Two-Cycle Target Labeling protocol is followed as suggested by the manufacturer and described succinctly as follows and shown graphically in the figure at the end of this Materials and Methods section: Total RNA (100 ng/uL) is retro-transcribed using T7-Oligo(dT) Promoter primers in the synthesis reaction of the first complementary DNA chain (cDNA). After treatment with RNAase H, the second cDNA chain is synthesized, which will serve as template in the Transcription reaction in vitro (TVI). The first TVI reaction is carried out with T7 polymerase RNA and unmarked ribonucleotides for the amplification of complementary RNA (cRNA). These cRNAs are retro-transcribed in the synthesis step of the first cDNA chain of the second cycle using random primers. Subsequently, T7-Oligo(dT)-Promoter primers are employed for the synthesis of the second chain of cDNA, generating the double-helix cDNA template that contains the promoter T7 sequence. This cDNA is amplified and marked in a second TVI reaction using the T7 polymerase DNA and a mixture of ribonucleotides/biotinylated nucleotide analog. These target biotinylated cDNAs are cleaned, fragmented, and hybridized to the GeneChip® expression microarrays. After hybridization, fluorescent marking was performed with a streptavidin-phycoerythrin and biotinylated anti-streptavidin antibody amplifier system. Fluorescence is detected with a high-resolution laser scanner.Reading and Analysis of Expression Microarrays:We will utilize the Expression Console of Affymetrix software to evaluate the quality of the microarrays and will correct the background signal with standard methods [49,50]. For signal intensity-level normalization, we will employ "non-supervised" methods, which use the data of all of the experiment's microarrays; this will allow us to render these comparable among themselves, because what a microarray assay evaluates is gene expression by means of fluorescence intensities; thus, it is important to establish cut-off points from which we can consider under- or overexpression. Once the data are normalized, the final stage is to resume the values of all the probes that exist for each gene in the microarray in a sole value, which is the gene's expression level. For detection of differentially expressed genes, we will construct a linear model that includes all of the experiment's microarrays simultaneously; in this manner, we will be able to analyze contrasts between group A (patients with metastasis to CNS during the follow-up period) and group B (patients without metastasis to CNS during the same period). As internal control, we will prove the differential expression of some genes by RT-PCR in real time. Results will be represented in blocks of heat maps and in tables, in which the most active genes are listed along with their functional description. For risk-profile validation, we will perform leave-one-out cross validation method and will postulate a second cohort for this objective.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* With auto-sufficiency
* Biopsy procedure approved
* Any TNM status
* Consulting at the National Institutes of Cancerology or Respiratory Diseases
* Informed consent signed

Exclusion Criteria:

* Comorbidity with other cancer type, hereditary or autoimmune diseases and treatment with immunosuppressor drugs
* Previous treatment with adjuvant or neoadjuvant chemo- or radiotherapy
* No specimen availability
* No diagnosis of non-small-cell lung cancer at histopathology sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed or suggested diagnosis of non-small-cell lung cancer, consulting at the National Institutes of Cancerology or Respiratory Diseases (INCan, INER; Mexico City, Mexico)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Central nervous system metastasis development | 8 months

SECONDARY OUTCOMES:
Death | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: David Saavedra-Pérez, MD, Principal Investigator — Instituto Nacional de Cancerologia de Mexico; Oscar Arrieta, MD, Study Chair — Instituto Nacional de Cancerologia de Mexico; Enrique Guzmán, MD, Study Director — Instituto Nacional de Enfermedades Respiratorias; Gabriela Mercado, MSc, Study Director — Instituto Nacional de Medicina Genómica; Elena Aréchaga, PhD, Study Director — Instituto Nacional de Cancerologia de Mexico; Claudia González, PhD, Study Director — Metropolitan Autonomous University; Digna Pachuca, MD, Study Director — Instituto Nacional de Cancerologia de Mexico
Locations (2):
- Mexico (2):
  - Instituto Nacional de Cancerología, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias, Mexico City